CLINICAL TRIAL: NCT05744661
Title: Effectiveness of Mechanical vs. Chemomechanical Methods in Removing Intracanal Calcium Hydroxide Medication: a Randomised Trial
Brief Title: Mechanical Vs Chemomechanical Method For Calcium Hydroxide Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, NEHAL AMIR, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PakistanIMS
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Necrotic Pulp; Chronic Apical Periodontitis
Keywords: Mechanical Method; Chemomechanical Method; Calcium Hydroxide; Intracanal Medicament
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: This is a Parallel type, Non-random Consecutive Sampling Technique. Patients reporting to the Department of Operative Dentistry & Endodontics, School of Dentistry with Necrotic teeth will be filtered. All participants who fulfil the Inclusion and Exclusion criteria will be enrolled in this study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a triple-blinded study. Participants will be unaware of the intervention they will recieve. All interventions will be performed by Single Care Provider (Clinician). Due to the nature of intervention, care provider cannot be masked. Data collector (Investigator) and Data Analyst(Outcome Assessor) both will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Mechanical Method) (Experimental): In Group A, Calcium Hydroxide Intracanal Medicament will be removed by using Mechanical Method in which Rotary Master Apical File will be used .
  Interventions: Other: Mechanical Method
- Group B ( Chemomechanical Method) (Experimental): In Group B, Calcium Hydroxide Intracanal Medicament will be removed by using Chemomechanical Method which involves Sonic Agitation of Endodontic irrigants.
  Interventions: Other: Chemomechanical Method

INTERVENTIONS:
Other: Mechanical Method — Use of Rotary Master Apical file for the removal of Calcium Hydroxide Medicament from Root Canal System
  Arms: Group A (Mechanical Method)
Other: Chemomechanical Method — Sonic Activation of Endodontic irrigants for the removal of Calcium Hydroxide from Root Canal System
  Arms: Group B ( Chemomechanical Method)

SUMMARY:
Type of study: Randomised Clinical trial To compare the effectiveness of Mechanical and Chemomechanical methods in the removal of Water-based Calcium hydroxide medicament from endodontic system.

Participants allocated in group A and B should be appointed for Endodontic treatment of Single rooted teeth diagnosed with Necrotic Pulp and Chronic Apical Periodontitis.

In group A, Calcium hydroxide medicament will be removed by using Mechanical method while in group B, Calcium hydroxide will be removed by using Chemomechanical method.

DETAILED DESCRIPTION:
This study is aimed at comparing the effectiveness of Mechanical and Chemomechanical methods for removal of Intracanal medication. Water-based Calcium hydroxide is used as an Intracanal medicament in this study. Participants aged 18 years and above presenting to the Outpatient department of Operative dentistry and Endodontics, School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad diagnosed with Necrotic Pulp with Chronic Apical Periodontitis will be randomly allocated in two groups A and B. On first visit, Root canal treatment will be initiated under rubber dam isolation. After locating canals, periapical radiograph for the working length will be taken. After working length has been confirmed, canal preparation will be done using Rotary file system. After canal has been prepared till working length, intracanal medicament is placed using Lentulospiral. Patient is recalled after 2 weeks. On next visit, Calcium hydroxide medicament will be removed by Mechanical method from group A. Mechanical method involves the use of Rotary file system for removal of medicament. In group B, Calcium hydroxide will be removed by using Chemomechanical method. Chemomechanical method involves the use of Sonic or Ultrasonic activation of irrigants for removal of medicament. After the removal of intracanal medicament, Periodical radiograph will be taken. Data will be taken on proforma and evaluation will be done for the effective removal of calcium hydroxide using a 4- point scoring system.

ELIGIBILITY:
Inclusion Criteria:

* SINGLE-ROOTED MAXILLARY AND MANDIBULAR TEETH
* NECROTIC TEETH WITH CHRONIC APICAL PERIODONTITIS
* STRAIGHT TO MODERATELY CURVED ROOT CANALS

Exclusion Criteria:

* PATIENTS WITH SYSTEMIC DISEASE
* PREGNANT AND IMMUNOCOMPROMISED PATIENTS
* TEETH WITH COMPROMISED PERIODONTAL HEALTH
* TEETH UNABLE TO BE RESTORED OR ISOLATED BY RUBBERDAM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Effective removal of Water-based Calcium hydroxide Intracanal medicament | Two week
  The effectiveness of mechanical and chemomechanical methods for the removal of calcium hydroxide will be evaluated using a 4 graded scoring system used in endodontics.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Amir, BDS, Principal Investigator — Pakistan Institiute of Medical Sciences
Locations (1):
- School of Dentistry, Pakistan Institute of Medical Sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anis Motiwala M, Badar SB, Ghafoor R. Comparison of Two Different Methods in the Removal of Oil-Based Calcium Hydroxide From Root Canal System: A Triple-Blinded Randomised Clinical Trial. Eur Endod J. 2021 Mar;6(1):38-43. doi: 10.14744/eej.2020.78941. PMID 33907070
- [Derived] Amir N, Noor N. Effectiveness of mechanical vs. chemomechanical methods in removing intracanal calcium hydroxide medication: a randomised trial. J Pak Med Assoc. 2024 Oct;74(10):1749-1754. doi: 10.47391/JPMA.10990. PMID 39407365